CLINICAL TRIAL: NCT00649701
Title: Phase 1 Online Intervention to Reduce Sexual Risk Among Men Who Have Sex With Men
Brief Title: Novel Internet-Based Interventions to Reduce Sexual Risk Among Men Who Have Sex With Men
Acronym: 5Part
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Public Health Solutions (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sabina Hirshfield, PhD /Senior Research Scientist, Public Health Solutions
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CDC-URS PS000415
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Last update posted 2008-06-20 (Estimated); Status verified 2008-06

CONDITIONS: HIV Infections
Keywords: HIV; Internet; MSM; Condom Use; Disclosure
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (No Intervention)
- 2 (Experimental): Text-based webpage
  Interventions: Behavioral: Standard Text-Based Prevention Web Page
- 3 (Experimental): Talking about HIV video
  Interventions: Behavioral: Talking About HIV
- 4 (Experimental): The Morning After video
  Interventions: Behavioral: The Morning After
- 5 (Experimental): Both videos
  Interventions: Behavioral: Both Videos

INTERVENTIONS:
Behavioral: Standard Text-Based Prevention Web Page — A link to the CDC.gov web page which describes HIV prevention among men who have sex with men.
  Arms: 2
Behavioral: The Morning After — A dramatic video about 4 gay men addressing sexual risk reduction within the context of alcohol use.
  Arms: 4
Behavioral: Talking About HIV — A documentary video addressing HIV disclosure, HIV testing, and condom use with the sub-context of drug use.
  Arms: 3
Behavioral: Both Videos — Morning After and Talking About HIV videos
  Arms: 5

SUMMARY:
The purpose of this study is to develop and test the efficacy of online HIV risk reduction interventions among men who have sex with men.

DETAILED DESCRIPTION:
This is an Internet-based, five-branch randomized controlled intervention, enrolling 3,000 adult MSM. The five branches include 1) a control condition receiving no intervention content, 2) a standard text-based prevention webpage, 3) an 8 minute dramatic video addressing sexual risk reduction within the context of alcohol use, 4) a 5 minute documentary video addressing HIV disclosure, HIV testing, and condom use with the sub-context of drug use, and 5) both videos. After completing the baseline survey, eligible participants who consent to participate in the intervention will be randomly assigned to the control condition or one of the four intervention conditions. The control condition will not include the delivery of any intervention content. All participants (branches 1-5) will be asked to complete a brief post-intervention survey (to measure intentions). All intervention participants will be invited to complete a final 60-day follow-up survey.

ELIGIBILITY:
Inclusion Criteria:

* Male;
* Age 18 and over;
* Ability to read and respond in English;
* Reside within the United States;
* Report oral or anal sex with any male (new partner or not) in the past 60 days AND report oral, anal or vaginal sex for the first time with any partner (male or female) in the past 60 days;
* Complete baseline survey
* Provide an email address;

Exclusion Criteria:

* Women and transgender persons

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3097 (Actual)
Dates: Start 2008-04; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
HIV disclosure, HIV testing, and condom use | 60 days

SECONDARY OUTCOMES:
drug and/or alcohol use before sex, and depressive and/or anxiety symptomatology (past 2 weeks) | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Sabina Hirshfield, PhD, Principal Investigator — Public Health Solutions
Locations (1):
- Public Health Solutions, New York, New York, United States

REFERENCES:
- [Derived] Hirshfield S, Chiasson MA, Joseph H, Scheinmann R, Johnson WD, Remien RH, Shaw FS, Emmons R, Yu G, Margolis AD. An online randomized controlled trial evaluating HIV prevention digital media interventions for men who have sex with men. PLoS One. 2012;7(10):e46252. doi: 10.1371/journal.pone.0046252. Epub 2012 Oct 2. PMID 23071551